CLINICAL TRIAL: NCT06785714
Title: Colorectal Cancer Screening in Xinxiang City
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Collaborators: Xinxiang Municipal Health Commission (Unknown); Xinxiang Center for Disease Control and Prevention (Unknown); Xinxiang Central Hospital (Other); The Affiliated People's Hospital of Xinxiang Medical University (Unknown); The Third Affiliated Hospital of Xinxiang Medical College (Unknown); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Chase 008
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual stool samples will be used to develop and evaluate the performance of biomarker assays to detect cancers and advanced precancerous lesions. Samples may be stored for up to 20 years. These stool samples will be deidentified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study is to evaluate the sensitivity of the fecal protein dual-index test reagent for the detection of colorectal cancer (CRC).

DETAILED DESCRIPTION:
The project uses fecal hemoglobin and transferrin dual-index combined with reagents that can be self-tested at home (referred to as fecal protein dual-index detection reagents), combined with colorectal cancer risk factor questionnaires, to carry out colorectal cancer screening in people of specific ages in the city, aiming to achieve early screening, early diagnosis and early treatment, and evaluate the effect of fecal protein dual-index detection reagents in early screening of colorectal cancer, so as to provide a scientific basis for optimizing the national screening program.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-74 years at time of consent
2. Have not had gastrointestinal resection

Exclusion Criteria:

1. Previous history of colorectal cancer
2. Patients who have been confirmed to have other malignant neoplastic diseases of the digestive system
3. Patients with severe heart, brain, lung disease or liver and kidney dysfunction or insufficiency
4. Those with severe mental disorders and language communication disorders
5. History of contraindications to colonoscopy
6. Pregnant women

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single cohort of patients aged between 45 and 84, with no known high risk features, undergoing routine colorectal cancer screening as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of colorectal cancer detection | 180 days
  Sensitivity of colorectal cancer detection
Specificity of advanced neoplasia detection | 180 days
  Specificity of advanced neoplasia detection

SECONDARY OUTCOMES:
Positive predictive value of colorectal cancer detection | 180 days
  Positive predictive value of colorectal cancer detection
Negative predictive value of colorectal cancer detection | 180 days
  Negative predictive value of colorectal cancer detection
Sensitivity and specificity of advanced adenoma detection | 180 days
  Sensitivity and specificity of advanced adenoma detection

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China